CLINICAL TRIAL: NCT04175860
Title: Design and Evaluation of Adherence to the Transition-discharge-hospital Plan in Patient-family Caregiver With Chronic Pathology in a Health Institution of the Metropolitan Area of Bucaramanga
Brief Title: Adherence to the Transition-discharge-hospital Plan in Patient-family Caregiver With Chronic Pathology
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Universidad de Santander (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: CIF 0314-19
Record Dates: First submitted 2019-11-21; First posted 2019-11-25 (Actual); Last update posted 2019-11-25 (Actual); Status verified 2019-11

CONDITIONS: Treatment Adherence and Compliance
MeSH Terms: conditions — Treatment Adherence and Compliance

STUDY DESIGN:
Intervention Model Description: Allocation: Randomized Endpoint Classification: Efficacy Study Intervention Model: Parallel Assignment
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): Consists of a series of non-pharmacological preventive interventions that will focus on the - transition-discharge-hospital program including individualized non-pharmacological interventions such as dyad characterization, competency assessment, risk assessment, inherent program strategies, and monitoring.
  The intervention or program " Hospital Discharge Plan" to develop was proposed by the Group of Chronic Care Patient and Family School of Nursing at the National University of Colombia. This program includes an educational session and weekly telephone follow-up according to the patient's risk characterization.
  Interventions: Behavioral: The intervention with the patient (Chronic Patient Care Group and his family.)
- Control group (No Intervention): This group of patients-family caregivers will be carried out the discharge activities that are regularly developed in the second level institution and recorded in a check-sheet and field diary.

INTERVENTIONS:
Behavioral: The intervention with the patient (Chronic Patient Care Group and his family.) — * Characterization: through the application of the characterization survey of the dyad (patient-caregiver),
  * Evaluation of the competence to care at home: Application of the instrument 'competence to care at home, long and short version both the patient and the family caregiver.
  * Risk assessment: this step is made based on the complexity of the treatment and the results of the evaluation the competence to care at home.
  Arms: Intervention group

SUMMARY:
To evaluate the therapeutic adherence of the patient-family caregiver with non-communicable chronic disease through the hospital transition-discharge plan program in a second level institution in the metropolitan area of Bucaramanga. Methods: The study will be a randomized controlled clinical trial in 100 participants who meet the inclusion criteria, distributed in a 1: 1 ratio for the intervention group and the control group, considering a confidence level of 90%, power of 80% and a reduction of 30%. Expected results: demonstrate the relevance of the program in the target population through the formation of information mechanisms between the parties involved in direct care, the development of skills and safety at home; the timely identification of the risks inherent to clinical conditions or possible complications associated with care, which aim to reduce the burdens related to the health - disease experience; also emphasize the continuity of the treatment established. On the other hand, achieve a more informed professional performance, prepared, transparent, that responds to the needs and expectations of the user in terms of monitoring and comprehensive therapeutic management. Impact: It is expected that this research will be the basis for the protocolization and implementation of the hospital discharge transition plan program in the health institution and subsequently develop a prospective study on a larger scale, which will allow evaluating its impact on the target population in order to reduce the complications, re-admissions and costs derived from the care of chronic patients.

DETAILED DESCRIPTION:
Noncommunicable chronic diseases are pathologies that over time require skills in the patient and family caregiver; to ensure safe and continuous care once they are discharged from health institutions. The approach of them represents multiple challenges in need of greater communication and education; for this, the importance of generating strategies through different interventions must be taken into account.

In this order of ideas, the program Plan of discharge or discharge consists of a coordinated intervention and executed by nursing staff that captures the patient dyad with chronic illness-family caregiver from his admission, stay and hospital discharge. The previous approach consists of a systematized guide that contemplates the following activities: 1) assessment of the family caregiver patient dyad to define the competence for care in the home (CARING), the level of risk and complexity of the care associated with the treatment in the home, according to defined risk: polypharmacy, parenteral medications, control medications and / or invasive devices; 2) education and instruction to the patient and the family caregiver during the hospital stay, anticipating the care needs at the time of discharge, with delivery of booklets, brochures and instructions, and 3) telephone follow-up for up to one month, by means of a 2-call call. week. (Melo Melo, Vargas Hernández, Carrrillo, & Alarcón Trujillo, 2017).

In a study carried out by (Sanchez, Carrillo Gonzalez, & Barrera, 2014) they refer that there exists a great variety of literature on the plan of transition and hospital discharge, in which it is possible to evidence a heterogeneous level opposite to concrete guidelines, to advance these plans, although this management is recommended in benefit of the users since the evidence on the effectiveness of the development of plans of care, as fundamental part of the continuous, safe and integral care of the patients and their families is very limited.

The support of professionals, institutions and the health system must respond to these demands to ensure the right to quality care for the sick person and the support required by his or her family caregiver, as well as other factors that influence access, security, continuity, social support with the use of appropriate information and communication technology and the strengthening of capacities for self-management and competence for care. (Carrillo Gonzalez , Sanchez Herrera, Gomez, Carreño, & Chaparro Diaz, 2017).

It is important to highlight that in a study conducted by (Sara Gutiérrez 2014) its objective was to identify the way of educating both the patient and the family at the time of discharge, it was possible to identify that the nursing staff does not give education to patients of the instructions issued by the medical staff; patients and their caregivers do not understand the care received and therefore 86% do not comply with the latest indications as well as 50% of re-entries is given for not having understood or had education in front of the care and instructions given at the time of discharge of the patient. (Gutierrez Suarez & Freire, 2014).

Regarding Effectiveness of the egress or transition plan for safe, comprehensive and continuous care, a trend is shown that would allow recommending the hospital transition and discharge plan, to support continuity, facilitate change, specify the guideline, avoid complications and decrease avoidable cost in patients with chronic, non-communicable disease. (Gutierrez Suarez & Freire, 2014)

On the other hand (Ginarte Arias, 2001) comments that in the majority of cases the patient and / or caregiver is blamed in the adherence; However, 'it is suggested that public policies and the health system could be directly related to the cause of non-adherence to treatment.' (Ginarte Arias, 2001) In addition, the weaknesses of the Health System contribute to the problem.

To assess adherence, different instruments have been designed, the most appropriate for this study being the Therapeutic Adherence Scale: it contains three factors, each with seven items distributed as follows: Control over the intake of medicines and foods, Medical follow-up behavioral and self-efficacy. Adherence is measured as a percentage, with 100 patients adhering. In this order of ideas, this instrument allows the evaluation of adherence in chronic diseases, without being directed to a specific disease. On the other hand, the authors have concluded that this scale identifies behavioral characteristics of patients, which favor or not their adherence to treatment (Soria Trujano, Vega Valero, & Navas Quiroz, 2009).

Program of Transition - Discharge Hospital, is based on strategies that can reduce adherence to treatment being predictive and key factors among which are: 'lack of knowledge of the disease, the therapeutic regimen and the consequences of non-compliance by the patient; lack of an adequate relationship between the patient and the doctor, complexity and long duration of treatment, asymptomatic disease, inadequate follow-up or lack of an elaborate plan on the abandonment of the medication; presence of adverse effects, cost of medication and / or copayment, failure to attend medical appointments, presence of psychological problems such as depression or anxiety, beliefs and perceptions of the patient. The transition and hospital discharge program starts from the patient's admission to hospital. the institution and the medication and presence of cognitive difficulties '. (Dilla, Valladares, Lizán, & Sacristán, 2009)

This research proposal is in the context and is articulated with the Comprehensive Health Care Policy (PAIS), where it addresses the different actors of the Health System to intervene in the social determinants that promote the health of people with chronic diseases. . It also shows the importance of intervening in public health with programs that in a short period contribute in a concrete way to the operative component in the Model of Integral Health Care (MIAS). (Ministry of Health and Social Protection, 2016)

ELIGIBILITY:
Inclusion Criteria:

* Patient with chronic pathology hospitalized in a second level institution in Floridablanca.
* Patient resident in the metropolitan area of Bucaramanga
* Patients over 18 years of age
* Patient with diagnosis at least 6 months old

Exclusion Criteria:

* People with communication difficulties.
* Patients with a health condition that at the time of the interview does not allow them to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-11-30 (Estimated); Primary Completion 2020-11-30 (Estimated); Study Completion 2021-02-28 (Estimated)

PRIMARY OUTCOMES:
1. Adherence to treatment | within the first 30 days
  Scale of therapeutic adherence for patients with chronic diseases, based on explicit behaviors developed by Rocio Soria Trujano, Cynthia Zaira Vega Valero and Carlos Nava Quiroz of the Facultad de Estudios Superiores Iztacala UNAM. Mexico.

SECONDARY OUTCOMES:
1. Competence for care | within the first 30 days
  Caregiver's capacity for care 'developed by the Chronic Patient Care Group and its Family of the Faculty of Nursing of the Universidad Nacional of Colombia. This instrument was developed based on the NOC (Nursing Outcomes Classification) taxonomies related to the preparation for care by the patient with chronic disease and family caregiver.

CONTACTS AND LOCATIONS:
Overall Officials: María S Campos de Aldana, Msc, Principal Investigator — Universidad de Santander
Locations (1):
- ESE Hospital San Juan de Dios Floridablanca, Floridablanca, Santander Department, Colombia

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make IPD available.

REFERENCES:
- [Background] Carrillo-González, G. M., Barreto-Osorio, R. V., Arboleda, L. B., Gutiérrez-Lesmes, O. A., Melo, B. G., & Ortiz, V. T. (2015). Competencia para cuidar en el hogar de personas con enfermedad crónica y sus cuidadores en Colombia. Revista de la Facultad de Medicina, 63(4), 665-675.
- [Background] González, G. M. C., Herrera, B. S., Ramírez, O. J. G., Moreno, S. P. C., & Díaz, L. C. (2017). Metodología de implementación del "plan de egreso hospitalario" para personas con enfermedad crónica en Colombia. Revista Med de la Facultad de Medicina, 25(2), 55-62.
- [Background] Mabel Carrillo G, Sanchez Herrera B, Arias Rojas EM. Validation of an instrument to assess the homecare competency of the family caregiver of a person with chronic disease. Invest Educ Enferm. 2015 Dec;33(3):449-455. doi: 10.17533/udea.iee.v33n3a08. PMID 28569952
- [Background] Dilla T, Valladares A, Lizan L, Sacristan JA. [Treatment adherence and persistence: causes, consequences and improvement strategies]. Aten Primaria. 2009 Jun;41(6):342-8. doi: 10.1016/j.aprim.2008.09.031. Epub 2009 May 7. No abstract available. Spanish. PMID 19427071
- [Background] familia, G. d. (s.f.). Bogotá: Universidad Nacional de Colombia. Ginarte Arias, Y. (2001). La adherencia terapéutica. Revista Cubana de Medicina general Integral, 502-505.
- [Background] Gutierrez Suarez, S., & Freire, C. (2014). Plan de egreso del paciente en el cuidado de enfermeria: cumplimiento en pacientes del área de Medicina Interna del hospita Pablo Arturo Suarez. Chile: Universidad de las americas.
- [Background] Melo Melo BG, Vargas Hernandez Y, Carrillo GM, Alarcon Trujillo DK. Effect of the programme Plan de egreso on chronically ill patients and their family caregivers. Enferm Clin (Engl Ed). 2018 Jan-Feb;28(1):36-43. doi: 10.1016/j.enfcli.2017.09.006. Epub 2017 Nov 17. English, Spanish. PMID 29153438